CLINICAL TRIAL: NCT03918109
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2 Study of OTO-313 Given as a Single Intratympanic Injection in Subjects With Subjective Tinnitus
Brief Title: OTO-313 in Subjects With Subjective Tinnitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 313-201901
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Tinnitus, Subjective
Keywords: tinnitus, intratympanic injection, gacyclidine
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicenter
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTO-313 (Experimental)
  Interventions: Drug: OTO-313
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-313 — single intratympanic injection of gacyclidine
  Arms: OTO-313
Drug: Placebo — single intratympanic injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, plasma pharmacokinetics (PK), and exploratory efficacy of OTO-313 administered as an intratympanic injection for the treatment of subjective tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Subject has subjective unilateral tinnitus and is consistently aware of their tinnitus throughout much of the waking day.
* Subject is able to use the electronic diary to complete their daily tinnitus ratings
* Subject's tinnitus is likely of cochlear origin, e.g., associated with sensorineural hearing loss; acute hearing loss from noise trauma, barotrauma, or traumatic cochlear injury (acute acoustic trauma, blast trauma, middle ear surgery, inner ear barotrauma); age-related hearing loss; resolved otitis media; ototoxic drug exposure.
* Subject is willing to comply with the protocol and attend all study visits.

Exclusion Criteria:

* Subject has pulsatile tinnitus, tinnitus resulting from traumatic head or neck injury, or tinnitus resulting from a tumor or stroke.
* Subject is pregnant or lactating.
* Subject has other clinically significant illness, medical condition or medical history at Screening or Baseline (Day 1) that, in the Investigator's opinion, would likely reduce the safety of study participation or compliance with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - House Clinic, Los Angeles, California
  - California Head & Neck Specialists, San Diego, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Silverstein Institute/Ear Research Foundation, Sarasota, Florida
  - ChicagoENT, Chicago, Illinois
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - Northwell Health, Hearing & Speech Center, New Hyde Park, New York
  - Northwell Health at ENT and Allergy Associates, White Plains, New York
  - Charlotte Eye Ear Nose & Throat Associates, Charlotte, North Carolina
  - Piedmont Ear, Nose, and Throat Associates, Winston-Salem, North Carolina
  - Worldwide Clinical Trials, San Antonio, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - WVU Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Part A, a total of 8 subjects registered for this study at a single site and signed an informed consent. Subject needed to have subjective unilateral or bilateral tinnitus (ringing or noise in the ear when there was no external cause) and be consistently aware of their tinnitus throughout much of the waking day.
Pre-assignment Details: Part A and Part B were conducted as 2 separate studies under a single protocol.
Groups:
- Part A OTO-313: Subjects received an 0.11 mg OTO-313 via an injection through the eardrum (IT injection) of a 0.2 mL medium chain triglycerides solution.
- Part A Placebo: Subjects received an injection through the eardrum of 0.2 mL medium chain triglycerides.
- Part B OTO-313: Subjects received 0.32 mg OTO-313 via an injection through the eardrum of a 0.2 mL medium chain triglycerides solution.
- Part B Placebo: Subjects received an injection through the eardrum of a 0.2 mL medium chain triglycerides solution.
Period: Overall Study
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo
Started | 6 | 2 | 17 | 18
Completed | 6 | 2 | 15 | 16
Not Completed | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A OTO-313: Subjects received 0.11 mg OTO-313 via an injection through the eardrum of a 0.2 mL medium chain triglycerides solution.
- Part A Placebo; Part B Placebo: Subjects received an injection through the eardrum of a 0.2 mL medium chain triglycerides solution.
- Total: Total of all reporting groups
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo | Total
Number analyzed (Participants) | 6 | 2 | 15 | 16 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 9 | 12 | 26
  >=65 years | 3 | 0 | 6 | 4 | 13
Age, Continuous [Median (Full Range); unit: years] | 64.0 [54 to 68] | 57.0 [57 to 57] | 58.0 [31 to 74] | 55.0 [33 to 71] | 57.5 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 7 | 7 | 17
  Male | 3 | 2 | 8 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 2 | 14 | 14 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 15 | 16 | 39
Months Since Initial Onset of Tinnitus [Mean (Standard Deviation); unit: Months] | 95.8 (87.09) | 49.0 (16.42) | 4.5 (1.96) | 4.20 (1.62) | 38.38 (37.84)

OUTCOME MEASURES:

1. Primary Outcome: Audiometry - Pure Tone Average Done Over 1000, 2000 and 4000 Hertz (HZ)
Description: Mean Change from Baseline to End of Study (baseline to Day 29 [4 weeks after dosing](Part A) or baseline to Day 57 [8 weeks after dosing] (Part B)). in Pure Tone Average Hearing Thresholds; a negative change indicates improvement.
Time Frame: Up to end of study (Part A - Day 29 [4 weeks after dosing]), (Part B - Day 57 [8 weeks after dosing])
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo
Number analyzed (Participants) | 6 | 2 | 14 | 15
decibels | -0.3 (2.66) | 0.71 (2.5) | -0.8 (6.44) | 0.3 (6.95)

2. Primary Outcome: Otoscopic Examination - Presence of Perforation in the Treated Ear at the End of Study Visit (Day 29 [4 Weeks After Dosing] (Part A) or Day 57 [8 Weeks After Dosing] (Part B)).
Description: Ear examinations were done at every visit. One of the important safety endpoints was an observation of a perforation in the ear drum that did not heal properly after the injection.
Time Frame: Up to end of study (Part A - Day 29 [4 weeks after the injection], Part B - Day 57 [8 weeks after the injection])
Measure: Count of Participants; unit: Participants
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo
Number analyzed (Participants) | 6 | 2 | 14 | 15
Participants
  Perforation present: pinhole size | 0 | 0 | 0 | 0
  Perforation present: ≤25% tympanic membrane | 0 | 0 | 0 | 0
  Perforation present: >25% and ≤50% tympanic membrane | 0 | 0 | 0 | 0
  Perforation present: >50% tympanic membrane | 0 | 0 | 0 | 0
  Perforation not present | 6 | 2 | 14 | 15

3. Other Pre Specified Outcome: Change From Baseline in Tinnitus Functional Index (TFI)
Description: Validated, 25-item questionnaire; index score from 0 to 100; a negative change indicates improvement. The 25 items of the TFI represent 8 subscales covering multiple domains of tinnitus severity: 1) Intrusive, 2) Sense of Control, 3) Cognitive, 4) Sleep, 5) Auditory, 6) Relaxation, 7) Quality of Life, and 8) Emotional. Subjects answer each TFI question by rating their experience over the past week. Each subscale has 3 questions with a response ranging from 0 (best response) to 10 (worst response) in regard to the impact of tinnitus in these different aspects of the subject's life. The highest raw score would be 250 and the lowest would be 0. The raw score is then divided by the total number of valid answers and that in turn is multiplied by 10 to give an overall score range from 0-100, with 0 representing no impact of tinnitus on their daily life and 100 representing complete impact of tinnitus on their daily life.
Time Frame: Up to the End of Study Visit (Part A - Day 29 [4 weeks after the injection]), (Part B - Day 57 [8 weeks after injection])
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo
Number analyzed (Participants) | 6 | 2 | 14 | 15
score on a scale | -4.2 (10.68) | 4.0 (0.00) | -12.9 (25.21) | -4.3 (18.18)

4. Other Pre Specified Outcome: Patient Global Impression of Change (PGIC)
Description: Change in overall tinnitus status as perceived by the subject; this was a subject-reported outcome that evaluated the change in overall "global" tinnitus status as perceived by the subject. The subject was asked: "Since the beginning of the clinical study, how would you rate your tinnitus?".
  The beginning of the clinical study in this context was the time prior to investigational product administration. The 7 response categories (and point scores) for the PGIC are:
  * Very much improved = 3
  * Much improved = 2
  * Minimally improved = 1
  * Unchanged = 0
  * Minimally worse = -1
  * Much worse = -2
  * Very much worse = -3
Time Frame: Measured at the end of study visit (Part A - Day 29 [4 weeks after injection]), (Part B - Day 57 [8 weeks after injection]).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo
Number analyzed (Participants) | 6 | 2 | 15 | 16
Participants
  Very much improved | 0 | 0 | 3 | 0
  Much improved | 0 | 0 | 1 | 1
  Minimally improved | 1 | 0 | 2 | 3
  Unchanged | 3 | 2 | 5 | 10
  Minimally worse | 1 | 0 | 3 | 0
  Much worse | 0 | 0 | 0 | 2
  Very much worse | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Reported or observed during or after dosing with the study drug up until the end of study (Part A - Day 29; Part B - Day 57)
Arm/Group | Part A OTO-313 | Part A Placebo | Part B OTO-313 | Part B Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 1/17 | 0/18
Other Adverse Events (participants affected / at risk) | 2/6 | 1/2 | 5/17 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A OTO-313 (N=6) | Part A Placebo (N=2) | Part B OTO-313 (N=17) | Part B Placebo (N=18)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A OTO-313 (N=6) | Part A Placebo (N=2) | Part B OTO-313 (N=17) | Part B Placebo (N=18)
Injection Site Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pruritis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ear Discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT03918109/Prot_SAP_000.pdf